CLINICAL TRIAL: NCT04801394
Title: Retrospective Analysis on Large Incisional Hernia in High Risk Patients: the Innovative "Neo-peritoneum" Approach With a Composite Mesh
Brief Title: Retrospective Analysis on Large Incisional Hernia in High Risk Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Claudio Gambardella, Clinical Professor, University of Campania Luigi Vanvitelli
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Combined mesh
Record Dates: First submitted 2021-03-11; First posted 2021-03-17 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Incisional Hernia; Large Incisional Hernia
MeSH Terms: conditions — Incisional Hernia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mesh Group (Experimental): Patient with large incisional hernia treated with FLaPp® mesh as neoperineium
  Interventions: Procedure: hernioplastic and insertion of FLaPp® composite mesh

INTERVENTIONS:
Procedure: hernioplastic and insertion of FLaPp® composite mesh — After the reduction of the large incisional hernia, the polypropylene transparent film of this mesh (lower flap) was sutured to the margins of the residual peritoneum and posterior rectus sheath as a "neo-peritoneum"; the macroporous light polypropylene layer (upper flap) was then sutured circumferentially with full-thickness transabdominal stitches in the retromuscular space.

SUMMARY:
Large incisional hernia (LIH) is a challenging condition where the abdominal wall is hopelessly compromised. Nowadays the best treatment option in this particularly frail subset of patients is a major issue. The Auhtors proposed the clinical experience with an innovative approach with the composite Free Lateral Polypropylene prosthesis (FLaPp®) mesh fashioned as "neoperitoneum" analyzing its feasibility and short/medium term results.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic patients with midline Large incisional hernia

Exclusion Criteria:

* lateral incisional hernias
* collagen diseases
* patients who recently have undergone chemotherapy and/or radiation therapy
* patients with acquired immunodeficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2010-04-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Early surgical outcome of FLaPp® prosthesis classified according to Clavien Dindo Classification | one month
  evaluation of feasibility of FLaPp® prosthesis in patients affected by LIH by the assessment of postoperative morbidity classified according to Clavien Dindo Classification
Evaluation of pain after FLaPp® prosthesis | one month
  Evaluation of postoperative pain through Visual Analague Scale
Mortality after FLaPp® prosthesis | One month
  Rate of posoperative mortality after FLaPp® prosthesis

SECONDARY OUTCOMES:
incisional hernia recurrence at medium term | 36 months
  assessment of postoperative recurrence after 36 months evaluated with clinical outcpatient control and CT scan
Patients' satisfatcion after FLaPp® prosthesis | 36 months
  Evaluated through the so-called 36 items Short-Form health survey

IPD SHARING:
Plan to Share IPD: No